CLINICAL TRIAL: NCT04159272
Title: OPEN.MIND | Can MINDfulness Help Vulnerable Youngsters to Ride a Challenging Emotional Tandem? OPENing up to Positivity While Simultaneously Accepting Negative Feelings
Brief Title: Effects of Mindfulness Training on the Emotional Experience and (Non-) Acceptance of Emotions in Adolescents
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Prof. dr. Filip Raes (Other)
Responsible Party: Sponsor-Investigator, Prof. dr. Filip Raes, Professor, KU Leuven
Organization: KU Leuven (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: s62523; G049019N (Other Grant/Funding Number: Research Foundation - Flanders)
Record Dates: First submitted 2019-11-06; First posted 2019-11-12 (Actual); Last update posted 2022-09-28 (Actual); Status verified 2022-09

CONDITIONS: Emotional Stress
MeSH Terms: conditions — Stress, Psychological

STUDY DESIGN:
Intervention Model Description: The intervention (MT) group receives a Mindfulness Training (MT) for 8 weeks in school, during regular school hours. The participants in the control group answer the questionnaires and complete the experience sampling assessments at the same timepoints as the intervention group, and follow the regular school curriculum.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mindfulness Training (Experimental): The MT programme adheres to a standardized protocol developed from MBSR (Kabat-Zinn, 1990) and MBCT (Segal et al., 2012) manuals and is adjusted to an adolescent population. Adjustments are based on our ample experience with mindfulness and adolescents in different contexts. Key objectives are: (1) to increase awareness of one's present moment experience; (2) to teach an attitude of openness and acceptance (non-judging) toward one's experience. This accepting attitude changes the person's relationship with the experience, being a detached and non-reactive orientation. Participants learn to recognize entanglement with one's thoughts and emotions and there is an increased understanding of one's spontaneous reactions. If adolescents adopt these skills, their negative emotions and cognitions will no longer be reinforced, creating the opportunity to deal with problematic thoughts and feelings.
  Interventions: Behavioral: Mindfulness Training
- Control (No Intervention): Participants follow their regular course curriculum.

INTERVENTIONS:
Behavioral: Mindfulness Training — The programme consists of 8 90-min sessions held once a week for 8 consecutive weeks. Each session consists of guided experiential mindfulness exercises, sharing of experiences of these exercises, reflections in small groups, psycho-education, and review of home practices. An overview of the core elements in each session is given in Van der Gucht et al. (2017). The in-class MT programme will be supported with a mindfulness for adolescents smartphone application to support practice at home.
  The curriculum is available in an open source platform. The training is supported by the use of homework assignments and audio material. The programme has already been piloted and reviewed in an expert group of mindfulness trainers and scientists working with youth in mental health care (Van der Gucht et al., 2017) and in refugee centres (Van der Gucht et al., 2019). The MT will be delivered by certified trainers (>3 years of experience). During the trial they will receive regular supervision.
  Arms: Mindfulness Training

SUMMARY:
The epidemiological data are alarming. Emotional distress, and depression in particular, is highly prevalent in adolescents, it has multiple problematic consequences and, most alarming, it is on the rise. All too often, these symptoms persist and lead to long-term and severe psychiatric problems. Mindfulness training (MT) is expected to counter both the non-acceptance of negative emotions (underlying depressed (sad) mood, anxiety and stress) and the dampening of positive emotions (underlying anhedonia). Vulnerable youngsters typically do not accept their negative emotions (which paradoxically further increases negative emotions) and also dampen positive emotions, as long as there are negative emotions present: a catch-22. MT, as a low-threshold intervention, is expected to 'unlock' this catch-22 by teaching participants to become non-judgmentally aware of thoughts, feelings, and sensations, and increasing their capacity to replace automatic, habitual, and often judgmental reactions with more conscious and skillful responses. That way, MT is hypothesized to reduce depressed (sad) mood, anxiety and stress and to promote protective positive emotions. On top, MT is expected to foster a healthier discourse among youngsters on their emotional lives as an alternative to society's malignant discourse that denounces negative emotions and over-focuses on the pursuit of happiness, which now backfires on vulnerable youngsters.

The aim of the present study is to evaluate the effects of MT in adolescents on their experience of negative emotions (i.e. symptoms of stress, anxiety and depression), suppression/acceptance of negative emotions, symptoms of anhedonia (i.e. lack of pleasurable feelings), dampening of positive emotions, social expectancies towards the (non-)expression and (non-)experience of negative emotions, and on several secondary outcomes or endpoints (e.g., loneliness, repetitive negative thinking, self-compassion). Pairs of two classes will be recruited from schools in Flanders, Belgium, and all adolescents (>14 years of age) of these selected classes will be invited to participate. One class in each pair will be randomly assigned to an 8-week MT during regular school hours supported by a newly developed mindfulness app for adolescents, while the other class (control group) follows the regular school curriculum. Before randomization, post-intervention and 3 months after the intervention, participant's current experience of negative emotions, their level of suppression/acceptance of negative emotions, dampening, and anhedonia will be assessed using experience sampling methods and self-report questionnaires.

The investigators hypothesize that mindfulness can help youngsters in their school context to become more accepting of their emotions and, that this 'opening up' not only leads to less distress and anhedonia, but also to less toxic social pressure amongst peers in school not to feel and not to talk about negative emotions. That way, mindfulness can help foster a social climate that promotes a more balanced embracement of emotions which is likely beneficial for young people's well-being.

ELIGIBILITY:
Inclusion Criteria:

* The study is open to all adolescents (>14yrs) of participating school classes.
* They should understand and speak Dutch.
* Written informed consent (including informed consent from a parent for those <18yrs) after been informed on all aspects of the study.

Exclusion Criteria:

* Not applicable

Min Age: 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 450 (Actual)
Dates: Start 2019-11-04 (Actual); Primary Completion 2022-06-03 (Actual); Study Completion 2022-06-03 (Actual)

PRIMARY OUTCOMES:
Change in Emotional Distress | Before randomisation, the week after the intervention and 3 months after the intervention; 10 times/day over 4 consecutive days
  A 3-item visual analogue scale ranging from 0 to 100 with the anchors "not at all" and "very much" is used to measure feelings of anxiety, stress and depression in the present moment. The final score will be computed as the average of the individual items.
Change in (Non)Acceptance of Negative Emotions | Before randomisation, the week after the intervention and 3 months after the intervention; 10 times/day over 4 consecutive days
  A 2-item visual analogue scale ranging from 0 to 100 with the anchors "not at all" and "very much" assesses the acceptance and non-acceptance of negative emotions since the last beep. The final score will be computed as the average of the individual items.
Change in Anhedonia | Before randomisation, the week after the intervention and 3 months after the intervention; 10 times/day over 4 consecutive days
  A 3-item visual analogue scale ranging from 0 to 100 with the anchors "not at all" and "very much" measures aspects of anhedonia in the present moment. The final score will be computed as the average of the individual items.
Change in Dampening | Before randomisation, the week after the intervention and 3 months after the intervention; 10 times/day over 4 consecutive days
  A single item visual analogue scale ranging from 0 to 100 with the anchors "not at all" and "very much" is used to assess dampening of positive emotions since the last beep.
Change in Social expectancies towards the (non-) expression and (non-) experience of negative emotions | Before randomisation, the week after the intervention and 3 months after the intervention; 10 times/day over 4 consecutive days
  A single item visual analogue scale ranging from 0 to 100 with the anchors "not at all" and "very much" measures social expectancies towards the non-expression and non-experience of negative emotions since the last beep.

SECONDARY OUTCOMES:
Change in Social expectancies towards the (non-) expression and (non-) experience of positive emotions | Before randomisation, the week after the intervention and 3 months after the intervention
  A single item visual analogue scale ranging from 0 to 100 with the anchors "not at all" and "very much" assesses social expectancies towards the expression and experience of positive emotions since the last beep.
Change in Repetitive Negative Thinking (RNT) - worry | Before randomisation, the week after the intervention and 3 months after the intervention
  A single item visual analogue scale ranging from 0 to 100 with the anchors "not at all" and "very much" is used to measure worry since the last beep.
Change in Loneliness | Before randomisation, the week after the intervention and 3 months after the intervention
  A single item visual analogue scale ranging from 0 to 100 with the anchors "not at all" and "very much" assesses feeling of loneliness in the present moment.
Change in Pro-social behaviour | Before randomisation, the week after the intervention and 3 months after the intervention
  A single item visual analogue scale ranging from 0 to 100 with the anchors "not at all" and "very much" is used to assess pro-social behaviour since the last beep.
Change in Self-compassion | Before randomisation, the week after the intervention and 3 months after the intervention
  A single item visual analogue scale ranging from 0 to 100 with the anchors "not at all" and "very much" measures self-compassion since the last beep.
Change in the Depression Anxiety Stress Scales (DASS-21) | Before randomisation, the week after the intervention and 3 months after the intervention
  The DASS is a 21-item scale and is comprised of three sub-scales that measure symptoms of depression, anxiety and stress over the past week. Items are scored on a 4-point Likert scale ranging from "0" (did not apply to me at all) to "3" (applied to me very much or most of the time).
Change in the Leuven Anhedonia Self-report Scale (LASS) | Before randomisation, the week after the intervention and 3 months after the intervention
  The LASS is a 12-item scale designed to assess consummatory, anticipatory, and motivational aspects of anhedonia over the past two weeks. Items are scored on a 5-point Likert scale ranging from "1" (completely untrue) to "5" (completely true).
Change in the Dampening subscale of Responses to Positive Affect questionnaire (RPA) | Before randomisation, the week after the intervention and 3 months after the intervention
  The dampening subscale of the RPA is used to measure dampening responses to positive affective states using 6 items on a 4-point Likert scale ranging from "1"(almost never) to "4"(almost always).
Change in the Non-Acceptance and Suppression of Negative Emotions Scale (NASNES) | Before randomisation, the week after the intervention and 3 months after the intervention
  The NASNES is a 10-item scale designed to assess the extent of suppression vs. acceptance of negative emotions on a 7-point Likert scale ranging from "1"(not at all) to "7"(very much).
Change in the Adapted and extended Social Expectancies to experience Depression and Anxiety Scale (SEDAD) | Before randomisation, the week after the intervention and 3 months after the intervention
  The 26-item SEDAD was adapted to the class climate and extended to assess social expectancies about the (non-)experience and (non-)expression of positive thoughts and emotions on a 9-point Likert scale ranging from "1" (strongly disagree) to "9" (strongly agree).
Change in the Core Characteristics Subscale of the Perseverative Thinking Questionnaire (PTQ) | Before randomisation, the week after the intervention and 3 months after the intervention
  The core characteristics subscale of the PTQ measures the main characteristics of repetitive negative thinking, namely the repetitiveness, the intrusiveness and the difficulty of disengaging. Its 9 items are rated on a 5-point Likert scale ranging from "0" (never) to "4" (always).
Change in the Self-Compassion Scale - Short Form | Before randomisation, the week after the intervention and 3 months after the intervention
  The 12-item short form of the Self-Compassion Scale assesses the main components of self-compassion, namely self-kindness vs. self-judgment, common humanity vs. isolation and mindfulness vs. over-identification. Items are rated on a 5-point Likert scale ranging from "1" (almost never) to "5" (almost always).
Change in the UCLA Loneliness Scale | Before randomisation, the week after the intervention and 3 months after the intervention
  The 8-item Loneliness Scale measures participants' loneliness on a 5-point Likert scale ranging from "1" (completely disagree) to "5" (completely agree).
Change in the Prosocial behaviour subscale of the Prosocialness Scale | Before randomisation, the week after the intervention and 3 months after the intervention
  The Prosocialness Scale is comprised of different subscales including the prosocial behaviour subscale. Its 6-items are rated on a 5-point Likert scale ranging from "1" (never/ hardly ever true) to "5" (almost always/ always true).
Change in the Short Form of the Comprehensive Inventory of Mindfulness Experiences (CHIME-SF) | Before randomisation, the week after the intervention and 3 months after the intervention
  The 24-item CHIME-SF measures different mindfulness skills including awareness of internal experiences, awareness of external experiences, acting with awareness, accepting and non-judgmental attitude, nonreactive decentering, openness to experiences, awareness of thought's relativity, and insightful understanding using a 6-point Likert scale ranging from "1" (almost never) to "6" (almost always).
Change in the Paying Attention to Your Surroundings scale (PAYS) | Before randomisation, the week after the intervention and 3 months after the intervention
  The 13-item PAYS scale assesses participants' attention for their surroundings including nature and architecture on a 9-point Likert scale ranging from "1" (totally disagree) to "9" (totally agree).
Change in the Pro-Environmental Behaviour Scale (PEB) | Before randomisation, the week after the intervention and 3 months after the intervention
  The PEB is a 15-item scale and is comprised of four subscales: environmental citizenship, conservation, food and transportation. Its items are rated on a 4-point Likert scale ranging from "0" (never) to "3" (always).

CONTACTS AND LOCATIONS:
Overall Officials: Filip Raes, Prof dr., Principal Investigator — KU Leuven
Locations (11):
- Belgium (11):
  - GO! Atheneum Ekeren, Antwerp
  - GO! KA Antwerpen, Antwerp
  - Leiepoort campus Sint-Hendrik, Deinze
  - Go! Lyceum Gent, Ghent
  - Heilig-Hart&College Halle, Halle
  - GO! Atheneum Heist, Heist-op-den-Berg
  - KOBOS Secundaire scholen, Kapelle-op-den-Bos
  - Heilig-Hart Instituut Heverlee, Leuven
  - KA Merksem, Merksem
  - GO! atheneum Oudenaarde, Oudenaarde
  - Vita et Pax Schoten, Schoten

IPD SHARING:
Plan to Share IPD: Yes
Moderately sensitive information including age, demographic data, all other data coming from questionnaires and experience sampling data using smartphones will be pseudo-anonymized and shared.
Supporting Information: Study Protocol
Time Frame: The coded, pseudonomized dataset will be uploaded in a csv format to OSF (in a restricted access repository) upon publication of the research results.
Access Criteria: Coded, pseudonomized data can be shared with regulatory authorities, ethical committees, other parties that collaborate with the research team and will be shared, as mentioned above, on the OSF platform. Other researchers will only have access to the coded, pseudonomized data, and only if they agree with the confidentiality rules agreed upon within this study.

REFERENCES:
- [Background] Abela, J. R., & Hankin, B. L. (Eds.). (2008). Handbook of depression in children and adolescents. Guilford Press.
- [Background] Bastin M, Nelis S, Raes F, Vasey MW, Bijttebier P. Party Pooper or Life of the Party: Dampening and Enhancing of Positive Affect in a Peer Context. J Abnorm Child Psychol. 2018 Feb;46(2):399-414. doi: 10.1007/s10802-017-0296-3. PMID 28391490
- [Background] Bauer DJ, Preacher KJ, Gil KM. Conceptualizing and testing random indirect effects and moderated mediation in multilevel models: new procedures and recommendations. Psychol Methods. 2006 Jun;11(2):142-63. doi: 10.1037/1082-989X.11.2.142. PMID 16784335
- [Background] Benjamini, Y., & Hochberg, Y. (1995). Controlling the False Discovery Rate: A Practical and Powerful Approach to Multiple Testing. Journal of the Royal Statistical Society. Series B (Methodological), 57(1), 289-300.
- [Background] Bergomi, C., Tschacher, W., & Kupper, Z. (2014). Konstruktion und erste Validierung eines Fragebogens zur umfassenden Erfassung von Achtsamkeit. Diagnostica, 60, 111-125.doi: 10.1026/0012-1924/a000109.
- [Background] Caprara, G. V., Steca, P., Zelli, A., & Capanna, C. (2005). A new scale for measuring adults' prosocialness. European Journal of psychological assessment, 21(2), 77-89.
- [Background] Cladder-Micus, M.B., Verweij, H., van Ravesteijn, H. et al. Mindfulness (2019) 10: 1893. https://doi.org/10.1007/s12671-019-01125-7
- [Background] Crane RS, Brewer J, Feldman C, Kabat-Zinn J, Santorelli S, Williams JM, Kuyken W. What defines mindfulness-based programs? The warp and the weft. Psychol Med. 2017 Apr;47(6):990-999. doi: 10.1017/S0033291716003317. Epub 2016 Dec 29. PMID 28031068
- [Background] Csikszentmihalyi M, Larson R. Validity and reliability of the Experience-Sampling Method. J Nerv Ment Dis. 1987 Sep;175(9):526-36. doi: 10.1097/00005053-198709000-00004. PMID 3655778
- [Background] Dejonckheere E, Bastian B, Fried EI, Murphy SC, Kuppens P. Perceiving social pressure not to feel negative predicts depressive symptoms in daily life. Depress Anxiety. 2017 Sep;34(9):836-844. doi: 10.1002/da.22653. Epub 2017 May 12. PMID 28499066
- [Background] Ehring T, Zetsche U, Weidacker K, Wahl K, Schonfeld S, Ehlers A. The Perseverative Thinking Questionnaire (PTQ): validation of a content-independent measure of repetitive negative thinking. J Behav Ther Exp Psychiatry. 2011 Jun;42(2):225-32. doi: 10.1016/j.jbtep.2010.12.003. Epub 2010 Dec 21. PMID 21315886
- [Background] Gotink RA, Chu P, Busschbach JJ, Benson H, Fricchione GL, Hunink MG. Standardised mindfulness-based interventions in healthcare: an overview of systematic reviews and meta-analyses of RCTs. PLoS One. 2015 Apr 16;10(4):e0124344. doi: 10.1371/journal.pone.0124344. eCollection 2015. PMID 25881019 (Retraction: PMID 30978236 PLoS One. 2019 Apr 12;14(4):e0215608)
- [Background] Goyal M, Singh S, Sibinga EM, Gould NF, Rowland-Seymour A, Sharma R, Berger Z, Sleicher D, Maron DD, Shihab HM, Ranasinghe PD, Linn S, Saha S, Bass EB, Haythornthwaite JA. Meditation programs for psychological stress and well-being: a systematic review and meta-analysis. JAMA Intern Med. 2014 Mar;174(3):357-68. doi: 10.1001/jamainternmed.2013.13018. PMID 24395196
- [Background] Hofmann SG, Sawyer AT, Witt AA, Oh D. The effect of mindfulness-based therapy on anxiety and depression: A meta-analytic review. J Consult Clin Psychol. 2010 Apr;78(2):169-83. doi: 10.1037/a0018555. PMID 20350028
- [Background] Hox, J. J., Moerbeek, M., & van de Schoot, R. (2010). Multilevel analysis: Techniques and applications: Routledge.
- [Background] Kabat-Zinn, J. (1990). Full catastrophe living: How to cope with stress, pain and illness using mindfulness meditation.New York: Delacorte.
- [Background] Kabat-Zinn, Jon. 1994. Wherever you go, there you are: mindfulness meditation in everyday life. New York: Hyperion.
- [Background] Khoury B, Lecomte T, Fortin G, Masse M, Therien P, Bouchard V, Chapleau MA, Paquin K, Hofmann SG. Mindfulness-based therapy: a comprehensive meta-analysis. Clin Psychol Rev. 2013 Aug;33(6):763-71. doi: 10.1016/j.cpr.2013.05.005. Epub 2013 Jun 7. PMID 23796855
- [Background] Luberto CM, White C, Sears RW, Cotton S. Integrative medicine for treating depression: an update on the latest evidence. Curr Psychiatry Rep. 2013 Sep;15(9):391. doi: 10.1007/s11920-013-0391-2. PMID 23943471
- [Background] Mathieu JE, Aguinis H, Culpepper SA, Chen G. Understanding and estimating the power to detect cross-level interaction effects in multilevel modeling. J Appl Psychol. 2012 Sep;97(5):951-66. doi: 10.1037/a0028380. Epub 2012 May 14. PMID 22582726
- [Background] Maynard, B. R., Solis, M. R., Miller, V. L., & Brendel, K. E. (2017). Mindfulness-Based Interventions for Improving Cognition, Academic Achievement, Behavior, and Socioemotional Functioning of Primary and Secondary School Students. Campbell Systematic Reviews 2017: 5. Campbell Collaboration.
- [Background] McGuirk L, Kuppens P, Kingston R, Bastian B. Does a culture of happiness increase rumination over failure? Emotion. 2018 Aug;18(5):755-764. doi: 10.1037/emo0000322. Epub 2017 Jul 17. PMID 28714701
- [Background] Merikangas KR, He JP, Burstein M, Swanson SA, Avenevoli S, Cui L, Benjet C, Georgiades K, Swendsen J. Lifetime prevalence of mental disorders in U.S. adolescents: results from the National Comorbidity Survey Replication--Adolescent Supplement (NCS-A). J Am Acad Child Adolesc Psychiatry. 2010 Oct;49(10):980-9. doi: 10.1016/j.jaac.2010.05.017. Epub 2010 Jul 31. PMID 20855043
- [Background] Mojtabai R, Olfson M, Han B. National Trends in the Prevalence and Treatment of Depression in Adolescents and Young Adults. Pediatrics. 2016 Dec;138(6):e20161878. doi: 10.1542/peds.2016-1878. Epub 2016 Nov 14. PMID 27940701
- [Background] Neff, K. D. (2003). Self-Compassion: An Alternative Conceptualization of a Healthy Attitude Toward Oneself. Self and Identity, 2(2), 85-101. http://dx.doi.org/10.1080/15298860309032
- [Background] Raes, F., Griffith, J. W., Van der Gucht, K., & Williams, J. M. G. (2014). School-based prevention and reduction of depression in adolescents: A cluster-randomized controlled trial of a mindfulness group program. Mindfulness, 5(5), 477-486.
- [Background] Rudolph, K. D. (2009). Adolescent depression. In I. H. Gotlib & C. L. Hammen (Eds.), Handbook of depression (pp. 444-466). New York, NY, US: The Guilford Press.
- [Background] Raes In Prep (2019)
- [Background] Bastian et al. In Prep.
- [Background] Russell D, Peplau LA, Cutrona CE. The revised UCLA Loneliness Scale: concurrent and discriminant validity evidence. J Pers Soc Psychol. 1980 Sep;39(3):472-80. doi: 10.1037//0022-3514.39.3.472. PMID 7431205
- [Background] Scherbaum, C. A., & Ferreter, J. M. (2009). Estimating statistical power and required sample sizes for organizational research using multilevel modeling. Organizational Research Methods, 12(2), 347-367
- [Background] Segal, Zindel V.; Mark, J.; Williams, G.; Teasdale, John D. (2012) Mindfulness-based cognitive therapy for depression: A new approach to preventing relapse. New York, NY, US: The Guilford Press.
- [Background] Spijkerman MP, Pots WT, Bohlmeijer ET. Effectiveness of online mindfulness-based interventions in improving mental health: A review and meta-analysis of randomised controlled trials. Clin Psychol Rev. 2016 Apr;45:102-14. doi: 10.1016/j.cpr.2016.03.009. Epub 2016 Apr 1. PMID 27111302
- [Background] Van der Gucht K, Takano K, Raes F, Kuppens P. Processes of change in a school-based mindfulness programme: cognitive reactivity and self-coldness as mediators. Cogn Emot. 2018 May;32(3):658-665. doi: 10.1080/02699931.2017.1310716. Epub 2017 Mar 31. PMID 28361569
- [Background] Van der Gucht, K., Takano, K., Kuppens, P., & Raes, F. (2017). Potential Moderators of the Effects of School-Based Mindfulness Program on Symptoms of Depression in Adolescents. Mindfulness, 8 (3), 797-806.
- [Background] Van der Gucht K, Takano K, Labarque V, Vandenabeele K, Nolf N, Kuylen S, Cosyns V, Van Broeck N, Kuppens P, Raes F. A Mindfulness-Based Intervention for Adolescents and Young Adults After Cancer Treatment: Effects on Quality of Life, Emotional Distress, and Cognitive Vulnerability. J Adolesc Young Adult Oncol. 2017 Jun;6(2):307-317. doi: 10.1089/jayao.2016.0070. Epub 2016 Dec 21. PMID 28002681
- [Background] Van der Gucht K, Dejonckheere E, Erbas Y, Takano K, Vandemoortele M, Maex E, Raes F, Kuppens P. An experience sampling study examining the potential impact of a mindfulness-based intervention on emotion differentiation. Emotion. 2019 Feb;19(1):123-131. doi: 10.1037/emo0000406. Epub 2018 Mar 26. PMID 29578747
- [Background] Van der Gucht K., Glas J., De Haene L., Kuppens P., Raes F. (2019). A Mindfulness-Based Intervention for Unaccompanied Refugee Minors: A pilot study using mixed methods evaluation. Journal of Child and Family Studies, 28(4), 1084-1093.
- [Background] Vollestad J, Nielsen MB, Nielsen GH. Mindfulness- and acceptance-based interventions for anxiety disorders: a systematic review and meta-analysis. Br J Clin Psychol. 2012 Sep;51(3):239-60. doi: 10.1111/j.2044-8260.2011.02024.x. Epub 2011 Sep 9. PMID 22803933
- [Background] Whitmarsh, L., & O'Neill, S. (2010). Green identity, green living? The role of pro-environmental self-identity in determining consistency across diverse pro-environmental behaviours. Journal of Environmental Psychology, 30(3), 305-314.